CLINICAL TRIAL: NCT03128138
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Describe Pharmacokinetics/Pharmacodynamics, and the Safety and of SPH3127 Tablet in Chinese Healthy Volunteers
Brief Title: Single Ascending Dose Study of Safety and Tolerability of SPH3127 Tablet in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPH3127-101
Record Dates: First submitted 2017-01-05; First posted 2017-04-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2021-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — SPH3127

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25 mg SPH3127 tablet-Dose 1 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet, 25mg, po. 1 tablet.
  2 Volunteers, Single dose of Placebo tablet, 25mg, po. 1 tablet.
  Interventions: Drug: SPH3127
- 50 mg SPH3127 tablet-Dose 2 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet, 50mg, po. 1 tablet.
  2 Volunteers, Single dose of Placebo tablet, 50mg, po. 1 tablet.
  Interventions: Drug: SPH3127
- 100 mg SPH3127 tablet-Dose 3 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet, 100mg, po. 1 tablet.
  2 Volunteers, Single dose of Placebo tablet, 100mg, po. 1 tablet.
  Interventions: Drug: SPH3127
- 200 mg SPH3127 tablet-Dose 4 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet,100mg, po. 2 tablet.
  2 Volunteers, Single dose of Placebo tablet, 100mg, po. 2 tablet.
  Interventions: Drug: SPH3127
- 400 mg SPH3127 tablet-Dose 5 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet,100mg, po. 4 tablet.
  2 Volunteers, Single dose of Placebo tablet, 100mg, po. 4 tablet.
  Interventions: Drug: SPH3127
- 800 mg SPH3127 tablet-Dose 6 (Experimental): 6 Volunteers, Single dose of SPH3127 tablet,100mg, po. 8 tablet.
  2 Volunteers, Single dose of Placebo tablet, 100mg, po. 8 tablet.
  Interventions: Drug: SPH3127

INTERVENTIONS:
Drug: SPH3127 — Drug: SPH3127 Tablet
  Drug: Placebo Tablet

SUMMARY:
1. To evaluate safety, tolerability and pharmacokinetics (PK) and pharmacodynamics (PD) characteristics of SPH3127 dose escalation, a single oral dose in Chines healthy volunteers.
2. To explore the appropriate dose and provide the basis for the subsequent clinical trials.

DETAILED DESCRIPTION:
48 healthy volunteers will participate in this trial. Participants will be divided into 6 group, 25mg，50mg，100mg，200mg，400mg and 800mg. In each group, 6 participants will take SPH3127 tablet, while 2 participants will take placebo randomly. Safety data and PK/PD data will be collected as protocol described.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults,age >=18 years.Single gender should no less than a third of total subjects in each group.
* BMI should be18 to 24 kg/m2 (including threshold), allowing the lowest weight 50 kg (including threshold) for the male and 45 kg (including threshold) for the female.
* understand details of significance, benefit, inconvenience and potential danger of the research program, voluntarily signed informed consent.

Exclusion Criteria:

* during pregnancy, nursing mothers, and plans to test in the first 6 months (grant) pregnant;
* abnormal results in physical examination, laboratory examination and have clinical significance (such as: liver function examination - aspartate aminotransferase (AST)/alanine aminotransferase (ALT) is more than 1.5 times of the upper limit of normal).
* with cardiovascular, liver, kidney, gastrointestinal, nervous system, blood system and familial blood disease, thyroid dysfunction or abnormal mental illness;
* has a history of drug allergy and allergic constitution;
* took birth control pills within 6 weeks;
* used any drugs (including Chinese herbal medicine) within 1 week;
* participated in blood donation within 2 months ;
* participated in any drug clinical trials (as subjects) within three months;
* any positive result in virus serology check: human immunodeficiency virus antigen antibody (HIV Ag/Ab) 、hepatitis c virus (HCV) - IgG antibody to IgG, hepatitis b surface antigen (HBsAg) and treponema pallidum antibody (TP);
* addicted to cigarettes, alcohol, drink coffee, strong tea and drug abuse;
* researchers think that exists any unfavorable factors to participate in the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of safety parameters [adverse events, laboratory data, vital signs, and ECG] | 10 days
  adverse events, laboratory data, vital signs, and ECG et al.

SECONDARY OUTCOMES:
Assessment of PK parameter 1 [Cmax] | 2 days
  Peak plasma concentration (Cmax)
Assessment of PD parameter 1 [Inhibition of Renion Activity (%)] | 2 days
  Inhibition of Renion Activity (%)
Assessment of PD parameter 2 [Blood pressure (mmHg)] | 2 days
  Blood pressure (mmHg)
Assessment of PK parameter 2 [tmax] | 2 days
  time to peak plasma concentration (tmax)
Assessment of PK parameter 3 [AUC] | 2 days
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: HONG MIAO, Principal Investigator — Shanghai Pharmaceuticals Holding Co., Ltd
Locations (1):
- The capital medical university affiliated Beijing anzhen hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jing S, Xu R, Yang K, Liu W, Zhang L, Ke Y, Xia G, Lin Y. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SPH3127: A Phase I, Randomized, Double-Blind, Placebo-Controlled Trial. Clin Ther. 2021 Apr;43(4):735.e1-735.e14. doi: 10.1016/j.clinthera.2021.01.025. Epub 2021 Feb 27. PMID 33653620